CLINICAL TRIAL: NCT03499925
Title: Theory Construction and Effect of Intervention on Pregnant Women With Gestational Hypertension and Endocrine Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201801053RINB
Record Dates: First submitted 2018-03-28; First posted 2018-04-17 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Pregnancy-related Complications
Keywords: mental health; intervention; pregnancy-related complications
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Telephone consultation effectiveness and cognitive behaviors
  Interventions: Behavioral: cognitive behaviors; Behavioral: Telephone consultation
- Comparison Group (No Intervention): Routine product inspection

INTERVENTIONS:
Behavioral: cognitive behaviors — Telephone consultation effectiveness and cognitive behaviors
  Arms: Test Group
Behavioral: Telephone consultation — Telephone consultation effectiveness and cognitive behaviors
  Arms: Test Group

SUMMARY:
Few reports have addressed mental health for women with pregnancy complication over a prolonged time period. Meanwhile, the caring model with intervention for women who have pregnancy complication needs to be developed. The aims of this study are to (1) describe and compare the differences in health indicators during pre-pregnancy, pregnancy and 1 year postpartum; (2) develop the theoretical framework of relationship among health indicators during perinatal period; (3) develop a telephone follow-up and consultation program and examine its effect on women's resilience, depression, anxiety and quality of life. In the first stage, a prospective longitudinal investigation will be performed in women at pregnancy and postpartum. Women with pregnancy-related complications will be recruited. All participants will complete questionnaires that assess demographic characteristics, obstetric and birth history, depression, anxiety, resilience and quality of life. Participants who are in early, middle, late pregnancy, 3-5 days, 1st, 3rd, and 6th month and 1 year postpartum will be contacted to complete the questionnaires by mail or at study site clinics. The sample size was estimated by drop rates and power calculation. Approximately 380 women in early pregnancy will be recruited at a medical center in northern Taiwan. The first stage of this study will be conducted over a 3-year period. In the second stage, randomized control trial with single blind will be used to recruit eligible subjects from women in the waiting room for prenatal examination at a medical center in Taipei. The eligible subjects will be randomized into a control or experimental group. The women in the control group will receive usual care and those in the experimental group will receive four instances of telephone follow-up or face-to-face consultation. Two groups will receive 3 times measurements of depressive symptom, anxiety, resilience and quality of life. Meanwhile, Investigators will assess the health indicators of women's newborn. Data will be analyzed by independent t-test and generalized estimating equations. Forty-eight subjects will be recruited in each group. Totally, 300 subjects will be approached in terms of including a 30% dropout rate. The second stage of this study will be conducted over a 2-year period.

ELIGIBILITY:
Inclusion criteria

1. age less than or equal to 20
2. pregnancy less than 35 weeks
3. CES-D questionnaire score greater than or equal to 16 points or State-Trait Anxiety Inventory-State(STAI-S) questionnaire score greater than 40 points
4. Ability to speak Chinese or Taiwanese, or willing to use translation services to help complete questionnaires and interventions
5. Ability to complete follow-up visits and electronic surveys
6. Agree to participate in the study and sign the consent form

Exclusion criteria

1. People with chronic diseases or congenital diseases before pregnancy.
2. Women who are not scheduled to continue to undergo probation or production at the study site.
3. Those who have major mental illnesses and are unable to complete self-administered questionnaires.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2018-04-23 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
CES-D | one week
  The Center for Epidemiological Studies-Depression (CES-D) scale asked the subject how often depressive symptoms had occurred in the past week. There were four frequencies: no, very few (less than one day per week), sometimes (every Monday to two days), and frequent (three to seven days per week). Options To assess each symptom, score 0 to 3 for each question. After the forward question is scored backwards, the total score for the 20 questions is between 0 and 60. Radloff Radloff suggested that the results should be explained by the total score of the scale. The total score is suggested to be interpreted by the total score of the scale. The total score is recommended to be explained by the total score of the scale, and the total score is recommended to be explained by the total score of the scale. The higher the total score, the more severe the depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-Ru Chang, PHD, Principal Investigator — PHD
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan